CLINICAL TRIAL: NCT03153423
Title: Basic Intermittent Exotropia; is the Axial Length of the Globe One of the Prognostic Factors for Overcorrection and Undercorrection After Binocular Surgery
Brief Title: Basic Intermittent Exotropia and Risk Factors for Postoperative Overcorrection and Under Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Lecturer of ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia2017
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basic intermittent exotropia patients (Other)
  Interventions: Procedure: Strabismus surgery

INTERVENTIONS:
Procedure: Strabismus surgery — Recession and resection of horizontal extra ocular muscles

SUMMARY:
To evaluate preoperative risk factors for overcorrection and undercorrection following surgery for basic intermittent exotropia such as axial length of the globe, refractive error, age and sex

ELIGIBILITY:
Inclusion Criteria:

* Basic type intermittent exotropia

Exclusion Criteria:

* previous strabismus surgery restrictive strabismus

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Risk factors for postoperative overcorrections and under corrections | 6 months
  as axial length of the globe, age, sex and refractive error

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Ibrahiem, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of medicine - Minia University, Minya, Egypt